CLINICAL TRIAL: NCT00004128
Title: The Value of High Dose Versus Standard Dose ARA-C During Induction and of IL-2 After Intensive Consolidation/Autologous Stem Cell Transplantation in Patients (Age 15-60 Years) With Acute Myelogenous Leukemia. A Randomized Phase II Trial of the EORTC and the GIMEMA-ALWP
Brief Title: Combination Chemotherapy, Interleukin-2, and Peripheral Stem Cell Transplant in Treating Patients With Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067356; EORTC-06991; GIMEMA-EORTC-06991
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2008-04

CONDITIONS: Leukemia
Keywords: untreated adult acute myeloid leukemia; adult acute erythroid leukemia (M6); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute megakaryoblastic leukemia (M7); adult acute monocytic leukemia (M5b); adult acute minimally differentiated myeloid leukemia (M0); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22)
MeSH Terms: conditions — Leukemia; Leukemia, Erythroblastic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Megakaryoblastic, Acute; Congenital Abnormalities | interventions — aldesleukin; Filgrastim; Busulfan; Cyclophosphamide; Cytarabine; Daunorubicin; Etoposide; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: aldesleukin
Biological: filgrastim
Drug: busulfan
Drug: cyclophosphamide
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: etoposide
Procedure: autologous bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Giving combination chemotherapy before a peripheral blood stem cell transplant stops the growth of cancer cells by stopping them from dividing or killing them. After treatment, stem cells are collected from the patient's blood or bone marrow and stored. More chemotherapy or radiation therapy is given prepare the bone marrow for the stem cell transplant. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy and radiation therapy. Interleukin-2 may stimulate the patient's white blood cells to kill cancer cells.

PURPOSE: This randomized phase III trial is studying two different regimens of combination chemotherapy, interleukin-2, and peripheral stem cell transplant and comparing them to see how well they work in treating patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival rate in patients with acute myeloid leukemia treated with high-dose versus standard-dose cytarabine during induction.
* Compare the disease-free survival rate in patients treated with or without interleukin-2 following consolidation and autologous peripheral blood stem cell or bone marrow transplantation.
* Compare the feasibility of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients in the first randomization are stratified according to center, WBC (no greater than 25,000/mm^3 vs 25,000-99,000/mm^3 vs at least 100,000/mm^3), age (15 to 45 vs 46 to 60), and performance status (0-1 vs 2 vs 3). Patients in the second randomization are stratified according to center, first treatment arm (I vs II), number of induction courses to reach complete remission (CR), cytogenic/molecular genetic group at diagnosis (low vs high vs intermediate vs unknown), and autologous peripheral blood stem cell (PBSC) transplantation planned after consolidation (yes vs no).

First randomization

* Induction: Patients are randomized to 1 of 2 treatment arms:

  * Arm I: Patients receive standard-dose cytarabine IV over 24 hours on days 1-10, etoposide IV over 1 hour on days 1-5, and daunorubicin IV over 5 minutes on days 1, 3, and 5.
  * Arm II: Patients receive etoposide and daunorubicin as in arm I and high-dose cytarabine IV over 3 hours every 12 hours on days 1, 3, 5, and 7.
* Consolidation: When CR is reached, patients receive intermediate-dose cytarabine IV over 2 hours every 12 hours on days 1-6 and daunorubicin IV over 5 minutes prior to cytarabine on days 4, 5, and 6.
* Harvest: Patients who achieve CR and are ineligible for allogeneic PBSC transplantation receive filgrastim (G-CSF) subcutaneously (SQ) every 12 hours beginning 20 days after starting consolidation treatment and continuing until autologous PBSC are harvested. Autologous bone marrow is collected from patients with insufficient PBSC. Allogeneic PBSC are harvested for patients who have an HLA identical donor. Allogeneic bone marrow is harvested for high risk patients (under age 40) who have an unrelated bone marrow donor.
* Transplant preparative chemotherapy: It is recommended that patients receive cyclophosphamide on 2 consecutive days and total body irradiation on 3 days OR busulfan on days -8, -7, -6, and -5 followed by cyclophosphamide on days -4 and -3.
* Transplantation: PBSC or bone marrow is infused on day 0.

Second randomization

* Patients who achieve CR with full hematologic recovery but have no HLA identical donor are randomized to 1 of 2 treatment arms no earlier than day 22 after stem cell infusion.

  * Arm I: Patients receive interleukin-2 SQ once daily for 5 days. Treatment repeats every 4 weeks for 1 year in the absence of disease progression or unacceptable toxicity.
  * Arm II: Patients receive no further treatment. Patients are followed at 1, 4, and 13 months, then every 4 months for 3 years, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 2,000 patients (1,000 per treatment arm) will be accrued for the first randomization and a total of 577 patients (288 per treatment arm) will be accrued for the second randomization of this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* First randomization:

  * Untreated newly diagnosed acute myeloid leukemia (AML)
  * At least 30% blasts in bone marrow
  * All cytological types of AML except acute promyelocytic leukemia (M3)
  * No blast crisis of chronic myelogenous leukemia
  * No leukemias supervening after other myeloproliferative disease
  * No leukemias supervening after overt myelodysplastic disorders (e.g., refractory anemia with excess blasts) for more than 6 months duration
* Second randomization:

  * Must have achieved complete remission with full hematologic recovery following consolidation treatment
  * No HLA identical family donor
  * Not eligible for allograft
  * No high risk patient (under age 40) for whom an unrelated bone marrow donor has been found within 8 weeks of beginning consolidation treatment

PATIENT CHARACTERISTICS:

Age:

* 15 to 60

Performance status:

* WHO 0-3 (first randomization)
* WHO 0-2 (second randomization)

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 3 times upper limit of normal (ULN)

Renal:

* Creatinine no greater than 3 times ULN

Cardiovascular:

* No severe heart failure requiring diuretics
* Ejection fraction at least 50%

Other:

* First randomization:

  * No other progressive malignant disease except the following:

    * Secondary acute leukemias following curatively treated Hodgkin's disease (even if treated with anthracyclines)
    * Other curatively treated malignancies
    * Secondary leukemias following other exposure to alkylating agents or radiotherapy for other reason
  * No uncontrolled infection
  * No severe concurrent neurologic or psychiatric disease
  * No psychological, familial, sociological, or geographical condition that could preclude compliance
* Second randomization:

  * No nonmalignant systemic illness that would increase risk of participation in study
  * No uncontrolled infection
  * No other progressive malignant disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for AML except hydroxyurea
* Less than 7 days of prior hydroxyurea

Endocrine therapy:

* No more than 7 days of prior corticosteroid therapy for AML

Radiotherapy:

* No prior radiotherapy for AML

Surgery:

* Not specified

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2000 (Estimated)
Dates: Start 1999-09; Primary Completion 2008-01 (Estimated)

PRIMARY OUTCOMES:
Duration of overall survival and disease-free survival after first randomization
Duration of overall survival and disease-free survival after second randomization

SECONDARY OUTCOMES:
Response after induction and consolidation
Toxicity measured by Cancer and Leukemia Group B (CALGB) CTCAE v3.0 after induction and consolidation
Disease-free survival after complete remission (CR)
Disease-free interval from CR
Time to death in CR
Peripheral stem cell harvest after consolidation
Rate of completion of autologous peripheral blood stem cell transplantation (auto-PBSCT) and allogeneic stem cell transplantation (allo-SCT)

CONTACTS AND LOCATIONS:
Overall Officials: Roel Willemze, MD, PhD — Leiden University Medical Center; Giovanna Meloni, MD, Study Chair — University La Sapienza

REFERENCES:
- [Background] Maurillo L, Buccisano F, Spagnoli A, et al.: In acute myeloid leukemia, the use in induction of standard dose arac is associated with a better quality of response as compared to an induction regimen containing high dose arac. [Abstract] Blood 114 (22): A-1584, 2009.
- [Result] Aslanyan MG, Langemeijer SMC, Cilloni D, et al.: Incidence and clinical impact of TET2 mutations in acute myeloid leukemia patients treated within the EORTC/GIMEMA AML-12/06991 AML trial. [Abstract] Blood 114 (22): A-2609, 2009.
- [Result] Willemze R, Suciu S, Mandelli F, et al.: Value of low dose IL-2 as maintenance following consolidation treatment or autologous transplantation in acute myelogenous leukemia (AML) patients aged 15-60 years who reached CR after high dose (HD-AraC) vs standard dose (SD-AraC) cytosine arabinoside during induction: results of the AML-12 trial of EORTC and GIMEMA Leukemia Groups. [Abstract] Blood 114 (22): A-791, 2009.
- [Derived] Baron F, Stevens-Kroef M, Kicinski M, Meloni G, Muus P, Marie JP, Halkes CJM, Thomas X, Vrhovac R, Albano F, Lefrere F Sr, Sica S, Mancini M, Venditti A, Hagemeijer A, Jansen JH, Amadori S, de Witte T, Willemze R, Suciu S. Impact of induction regimen and allogeneic hematopoietic cell transplantation on outcome in younger adults with acute myeloid leukemia with a monosomal karyotype. Haematologica. 2019 Jun;104(6):1168-1175. doi: 10.3324/haematol.2018.204826. Epub 2018 Dec 6. PMID 30523055
- [Derived] Baron F, Stevens-Kroef M, Kicinski M, Meloni G, Muus P, Marie JP, Halkes CJM, Thomas X, Vrhovac R, Specchia G, Lefrere F Sr, Sica S, Mancini M, Venditti A, Hagemeijer A, Becker H, Jansen JH, Amadori S, de Witte T, Willemze R, Suciu S. Cytogenetic clonal heterogeneity is not an independent prognosis factor in 15-60-year-old AML patients: results on 1291 patients included in the EORTC/GIMEMA AML-10 and AML-12 trials. Ann Hematol. 2018 Oct;97(10):1785-1795. doi: 10.1007/s00277-018-3396-4. Epub 2018 Jun 20. PMID 29926156
- [Derived] Kroeze LI, Aslanyan MG, van Rooij A, Koorenhof-Scheele TN, Massop M, Carell T, Boezeman JB, Marie JP, Halkes CJ, de Witte T, Huls G, Suciu S, Wevers RA, van der Reijden BA, Jansen JH; EORTC Leukemia Group and GIMEMA. Characterization of acute myeloid leukemia based on levels of global hydroxymethylation. Blood. 2014 Aug 14;124(7):1110-8. doi: 10.1182/blood-2013-08-518514. Epub 2014 Jul 1. PMID 24986689
- [Derived] Willemze R, Suciu S, Meloni G, Labar B, Marie JP, Halkes CJ, Muus P, Mistrik M, Amadori S, Specchia G, Fabbiano F, Nobile F, Sborgia M, Camera A, Selleslag DL, Lefrere F Sr, Magro D, Sica S, Cantore N, Beksac M, Berneman Z, Thomas X, Melillo L, Guimaraes JE, Leoni P, Luppi M, Mitra ME, Bron D, Fillet G, Marijt EW, Venditti A, Hagemeijer A, Mancini M, Jansen J, Cilloni D, Meert L, Fazi P, Vignetti M, Trisolini SM, Mandelli F, de Witte T. High-dose cytarabine in induction treatment improves the outcome of adult patients younger than age 46 years with acute myeloid leukemia: results of the EORTC-GIMEMA AML-12 trial. J Clin Oncol. 2014 Jan 20;32(3):219-28. doi: 10.1200/JCO.2013.51.8571. Epub 2013 Dec 2. PMID 24297940